CLINICAL TRIAL: NCT04931186
Title: Retrospective Data Analysis of Patients Undergoing Lacrimal Drainage System Interventions at The Department of Ophthalmology and Optometry During The Years 2013 - 2017
Brief Title: Nasolacrimal Duct Obstruction
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Told, clinical Professor, Medical University of Vienna
Other Study IDs: NLDO 01309113
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Eye Diseases; Lacrimal Duct Obstruction
MeSH Terms: conditions — Eye Diseases; Lacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all patients
  Interventions: Other: retrospective analyis

INTERVENTIONS:
Other: retrospective analyis — retrospective analysis of data

SUMMARY:
1.1 Background Obstructions of the lacrimal drainage system can be differentiated based on anatomical location or severity. But also, differentiating between congenital and acquired nasolacrimal duct obstruction (NLDO) is possible. The incidence of congenital NLDO (CNLOD) has been shown to be approximately 20%. Most of the cases undergo spontaneous remission, as the ductus nasolacrimalis may open spontaneously. About 2-12% display a symptomatic course. 2. S: 290; 3; 4, 5 Acquired NLDO may occur during childhood and adulthood. The incidence of symptomatic acquired NLDO is around 30 cases per 100.000 people in an US-based cohort study. S: 293; 30 Two major anatomical closure sites have been described, which are on the one hand located at the between the punctum and canaliculus, and on the other hand located after the lacrimal sac. 1. S. ; 2. S: 293 1.2 Aim of this study The aim of this study is to assess the success rates for different types of primary tear duct surgery, performed from 2013 - 2017 at the department of Ophthalmology and Optometry, Medical University of Vienna.

Treatment success was defined as the absence of clinical signs of lacrimal drainage system obstruction (epiphora, increased tear leak, mucous discharge) and without the need for re-intervention.

It is further investigated whether the type of operation performed or whether the silicone tube used influence success rates.

1.3 Methods A retrospective chart analysis of all patients - independent of the underlying pathology - undergoing surgery of the lacrimal drainage system between 1st of January 2013 and 31st December 2017. Success rates and patient profiles will be analyzed not only for all patients, but also for subgroups based on the underlying pathology and operation performed.

ELIGIBILITY:
Inclusion criteria

* All charts of patients treated during the above-indicated period of time will be considered for this analysis.

Exclusion criteria

* incomplete medical records are considered an exclusion criterion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Charts of all patients - independent of the underlying pathology - undergoing surgery of the lacrimal drainage system between 1st of January 2013 and 31st December 2017. We expect approximately 700 eyes of 500 patients.
Sampling Method: Non-Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Success rate of NLDO interventions | 1.1.2013 - 31.12.2017

SECONDARY OUTCOMES:
Success rate of different surgical approaches | 1.1.2013 - 31.12.2017

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided